CLINICAL TRIAL: NCT02286739
Title: Prospective Clinical Study Evaluating Tibiofemoral Rotational Alignment Using Intraoperative Sensing During Total Knee Arthroplasty
Brief Title: Prospective Clinical Study Evaluating Tibiofemoral Rotational Alignment Using Intraoperative Sensing During Total Knee Arthroplasty (TKA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expected enrollment and follow-up not met
Sponsor: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 102
Record Dates: First submitted 2014-10-31; First posted 2014-11-10 (Estimated); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis
Keywords: Total Knee Arthroplasty; Rotational Alignment; Intraoperative Sensors; Patient Outcomes; Soft Tissue Balance
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A TKA without VERASENSE (Sham Comparator): Patients who undergo primary posterior cruciate ligament (PCL)-retaining or - sacrificing TKA without the use of VERASENSE to guide rotational alignment and balance.
  Interventions: Procedure: TKA without "Verasense"
- Group B TKA with VERASENSE (Active Comparator): Patients who undergo primary PCL-retaining or - sacrificing TKA with the use of VERASENSE to guide rotational alignment and balance.
  Interventions: Device: TKA with "Verasense"

INTERVENTIONS:
Device: TKA with "Verasense" — VERASENSE replaces the standard tibial trial inserts and is embedded with microelectronics and sensors to provide surgeons with real-time knee kinetic data. The data is wirelessly transmitted to a graphic display (VERASENSE Knee Application), allowing surgeons to quantify and assess soft tissue intercompartmental loads throughout the range of motion. The VERASENSE sensor is not an investigational device. OrthoSensor, Inc., received FDA pre-market submission (510K) clearance in 2009. The indication for use is a tool for adjustment of the femoral knee implant to reduce instability from flexion gap asymmetry. The VERASENSE sensor is sterile and single patient use.
  Arms: Group B TKA with VERASENSE
Procedure: TKA without "Verasense" — TKA will be performed manually without the use of Verasense
  Arms: Group A TKA without VERASENSE

SUMMARY:
The objectives of the study are twofold: 1) Evaluate how intra-operative sensing may assist the surgeon with tibiofemoral rotational alignment by testing the precision and variability of setting tray rotation to the mid-third of the tibial tubercle. 2) Understand if patients with a combined axial rotation couple at the tibiofemoral joint and quantitative intercompartmental balance, achieved with the use of VERASENSE, exhibit less post-operative knee pain and improved clinical outcomes. Radiographic outcomes will also be assessed to measure post-operative alignment and to evaluate the prevalence and location of radiolucency and/or osteolysis.

DETAILED DESCRIPTION:
Hypothesis: TKA with VERASENSE results in a more reliable and precise option for establishing implant-to-implant congruency and joint balance leading to less knee pain, faster return to normal activities and higher patient satisfaction compared to TKA without VERASENSE.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the indications for use for Triathlon® Total Knee System using VERASENSE™
* Subject must be diagnosed with one or more of the following conditions
* osteoarthritis
* rheumatoid or other inflammatory arthritis
* post-traumatic arthritis
* Subject is likely to be available for all study visits
* Subject is able and willing to sign the informed consent and follow study procedures

Exclusion Criteria:

* Prior Total Knee Arthroplasty
* Avascular Necrosis
* Any knee surgery other than meniscectomy (can be arthroscopic or open)
* Ligament insufficiencies, prior surgeries such as anterior cruciate ligament (ACL) or PCL reconstructions, posterolateral reconstructions, osteotomies, tibia plateau fractures
* Ipsilateral foot/ankle and hip arthritis
* Range of motion less than 90°, flexion contracture greater than 20°
* Subject has a mental condition that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Any subjects meeting any contraindication criteria as identified in the locally approved labeling for the device should be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Golladay, MD, Principal Investigator — Virginia Commonwealth University
Locations (6):
- United States (6):
  - The Cleveland Clinic Foundation, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Illinois Bone & Joint Institute, Morton Grove, Illinois
  - NYU Hospital for Joint Diseases, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A TKA Without VERASENSE: patients who undergo primary Posterior Cruciate Ligament (PCL-retaining or - sacrificing TKA without the use of VERASENSE to guide rotational alignment and balance.
  TKA without "Verasense": TKA will be performed manually without the use of Verasense
- Group B TKA With VERASENSE: patients who undergo primary PCL-retaining or - sacrificing TKA with the use of VERASENSE to guide rotational alignment and balance.
  TKA with "Verasense": VERASENSE replaces the standard tibial trial inserts and is embedded with microelectronics and sensors to provide surgeons with real-time knee kinetic data. The data is wirelessly transmitted to a graphic display (VERASENSE Knee Application), allowing surgeons to quantify and assess soft tissue intercompartmental loads throughout the range of motion. The VERASENSE sensor is not an investigational device. OrthoSensor, Inc., received FDA 510K clearance in 2009. The indication for use is a tool for adjustment of the femoral knee implant to reduce instability from flexion gap asymmetry. The VERASENSE sensor is sterile and single patient use.
Period: Overall Study
Arm/Group | Group A TKA Without VERASENSE | Group B TKA With VERASENSE
Started | 170 | 162
Completed | 46 | 9
Not Completed | 124 | 153
Not completed — Verasense type posterior stabilizing (PS) | 37 | 16
Not completed — No Verasense type documented | 0 | 23
Not completed — Adverse Event | 1 | 2
Not completed — Lost to follow-up (LTFU), Patient withdrawal or Physician decision but not specified | 86 | 112

BASELINE CHARACTERISTICS:
Population: Baseline data was not collected for all participants.
Groups:
- Group A TKA Without VERASENSE: patients who undergo primary PCL-retaining or - sacrificing TKA without the use of VERASENSE to guide rotational alignment and balance.
  TKA without "Verasense": TKA will be performed manually without the use of Verasense
- Total: Total of all reporting groups
Arm/Group | Group A TKA Without VERASENSE | Group B TKA With VERASENSE | Total
Number analyzed (Participants) | 170 | 162 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Incomplete baseline data collected for all participants in each sub-category (Group A: 4 missing / Group B: 11 missing).
  years
    number analyzed (Participants) | 166 | 151 | 317
    (all) | 67.29 (8.42) | 68.06 (8.12) | 67.73 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Incomplete baseline data collected for all participants in each sub-category (Group A: 0 missing / Group B: 2 missing).
  Participants
    number analyzed (Participants) | 170 | 160 | 330
    Female | 112 | 101 | 213
    Male | 58 | 59 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Incomplete baseline data collected for all participants in each sub-category (Group A: 36 missing / Group B: 20 missing).
  Participants
    African American or Black: number analyzed (Participants) | 134 | 142 | 276
    African American or Black | 19 | 22 | 41
    Asian: number analyzed (Participants) | 134 | 142 | 276
    Asian | 0 | 3 | 3
    Hispanic or Latino: number analyzed (Participants) | 134 | 142 | 276
    Hispanic or Latino | 6 | 6 | 12
    Other: number analyzed (Participants) | 134 | 142 | 276
    Other | 4 | 2 | 6
    White: number analyzed (Participants) | 134 | 142 | 276
    White | 105 | 109 | 214
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg / m^2] — Population: Incomplete baseline data collected for all participants in each sub-category (Group A: 1 missing / Group B: 2 missing).
  kg / m^2
    number analyzed (Participants) | 169 | 160 | 329
    (all) | 31.29 (6.65) | 31.11 (6.27) | 31.20 (6.46)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Quantitatively Balanced and Unbalanced Knees in Primary Unilateral Total Knee Arthroplasty
Description: Evaluate how intra-operative sensing with VERASENSE may assist the surgeon with balancing.
  A load differential of up to 15 pound (lbs) or less between the medial and lateral condyles is indicative of soft-tissue balance. A load differential more than 15 lbs is indicative for soft-tissue unbalance.
Time Frame: Intra-operative with trial implants in place and after completing all surgical corrections.
Population: Data was not collected for all participants. Numbers analyzed represent evaluable cases.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A TKA Without VERASENSE | Group B TKA With VERASENSE
Number analyzed (Participants) | 133 | 123
Participants
  Participants with balanced knee | 65 | 103
  Participants with unbalanced knee | 68 | 20

2. Secondary Outcome: Knee Society Knee Scoring System
Description: "Patient Satisfaction" is a three-question 40-point scale and has a score of 0 (not satisfied) to 40 (very satisfied) that is collected preoperatively and at each follow-up visit.
  "Patient Expectations" is a five-question fifteen-point scale and has a score of 0 (low expectation) to 15 (high expectation) that is collected pre-operatively and post-operatively. The pre-operative questions reflect the patient's opinion on the extent to which the patient expects that the operation will improve their knee pain, and their ability to perform their activities of daily living and recreational activities. The post-operative questions reflect the extent to which the outcome after the operation has met the patient's pre-operative expectations with respect to pain and function.
  The "functional score" is composed of four subgroups (Walking and standing, standard activities, advanced activities, discretionary activities) and has a score of 0 (poor) to 100 (excellent).
Time Frame: pre-operative, 6 weeks, 6 months, 1 year, 2 years
Population: Data was not collected for all participants. Numbers analyzed represent evaluable cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A TKA Without VERASENSE | Group B TKA With VERASENSE
Number analyzed (Participants) | 165 | 140
units on a scale
  Satisfaction Score pre-operative | 13.61 (6.94) | 13.35 (6.85)
  Satisfaction Score 6 weeks: number analyzed (Participants) | 105 | 111
  Satisfaction Score 6 weeks | 26.20 (7.93) | 26.45 (8.28)
  Satisfaction Score 6 months: number analyzed (Participants) | 105 | 74
  Satisfaction Score 6 months | 31.11 (8.71) | 31.30 (8.93)
  Satisfaction Score 1 year: number analyzed (Participants) | 99 | 53
  Satisfaction Score 1 year | 32.44 (8.48) | 32.98 (8.22)
  Satisfaction Score 2 years: number analyzed (Participants) | 45 | 9
  Satisfaction Score 2 years | 32.15 (7.90) | 33.21 (7.32)
  Expectations Score pre-operative | 14.30 (1.40) | 14.19 (1.48)
  Expectations 6 weeks: number analyzed (Participants) | 105 | 111
  Expectations 6 weeks | 9.62 (2.72) | 9.50 (2.74)
  Expectations 6 months: number analyzed (Participants) | 105 | 74
  Expectations 6 months | 10.01 (2.82) | 9.92 (2.89)
  Expectations 1 year: number analyzed (Participants) | 99 | 53
  Expectations 1 year | 10.28 (3.08) | 10.44 (3.04)
  Expectations 2 years: number analyzed (Participants) | 45 | 9
  Expectations 2 years | 10.69 (3.35) | 10.81 (3.25)
  Functional Score pre-operative | 36.75 (15.88) | 37.13 (16.11)
  Functional Score 6 weeks 6 weeks: number analyzed (Participants) | 105 | 111
  Functional Score 6 weeks 6 weeks | 44.84 (19.02) | 46.73 (18.91)
  Functional Score 6 months: number analyzed (Participants) | 105 | 74
  Functional Score 6 months | 69.25 (19.24) | 68.95 (19.03)
  Functional Score 1 year: number analyzed (Participants) | 99 | 53
  Functional Score 1 year | 71.82 (17.34) | 72.44 (17.09)
  Functional Score 2 years: number analyzed (Participants) | 45 | 9
  Functional Score 2 years | 68.69 (18.65) | 69.77 (18.29)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the EuroQuol-5 Dimension Health Questionnaire (EQ-5D).
Description: The EQ-5D Time Trade-off (TTO) descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/comfort and anxiety/depression. Each dimension has three levels: no problems, some problems and extreme problems. The scores range from -0.59 (worst possible health state) to 1 (best possible health state).
Time Frame: Pre-operative, 6 weeks, 6 months, 1 year and 2 years
Population: Data was not collected for all participants. Numbers analyzed represent evaluable cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group A TKA Without VERASENSE: Patients who undergo primary PCL(posterior cruciate ligament)-retaining or - sacrificing TKA without the use of VERASENSE to guide rotational alignment and balance.
  TKA without "Verasense": TKA will be performed manually without the use of Verasense
Arm/Group | Group A TKA Without VERASENSE | Group B TKA With VERASENSE
Number analyzed (Participants) | 165 | 137
units on a scale
  EQ-5D TTO pre-operative | 0.66 (0.18) | 0.63 (0.19)
  EQ-5D TTO 6 weeks: number analyzed (Participants) | 118 | 111
  EQ-5D TTO 6 weeks | 0.75 (0.18) | 0.78 (0.15)
  EQ-5D TTO 6 months: number analyzed (Participants) | 107 | 74
  EQ-5D TTO 6 months | 0.87 (0.14) | 0.85 (0.16)
  EQ-5D TTO 1 year: number analyzed (Participants) | 98 | 52
  EQ-5D TTO 1 year | 0.86 (0.18) | 0.87 (0.13)
  EQ-5D TTO 2 years: number analyzed (Participants) | 46 | 9
  EQ-5D TTO 2 years | 0.86 (0.14) | 0.73 (0.18)

4. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The FJS is based on the patients' ability to forget about a joint as a result of the treatment. The FJS assessment is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
Time Frame: 6 weeks, 6 months, 1 year, 2 years
Population: Data was not collected for all participants. Numbers analyzed represent evaluable cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A TKA Without VERASENSE | Group B TKA With VERASENSE
Number analyzed (Participants) | 103 | 98
units on a scale
  FJS 6 weeks | 30.55 (25.52) | 33.31 (27.88)
  FJS 6 months: number analyzed (Participants) | 94 | 52
  FJS 6 months | 55.11 (26.89) | 55.46 (26.77)
  FJS 1 year: number analyzed (Participants) | 80 | 34
  FJS 1 year | 57.88 (28.23) | 60.34 (27.35)
  FJS 2 years: number analyzed (Participants) | 29 | 8
  FJS 2 years | 59.78 (32.22) | 65.73 (31.11)

ADVERSE EVENTS:
Time Frame: Date of inclusion to 2 years
Description: The definition of adverse event and/or serious adverse event does not differ from ClinicalTrilas.gov definition.
Arm/Group | Group A TKA Without VERASENSE | Group B TKA With VERASENSE
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/162
Serious Adverse Events (participants affected / at risk) | 8/170 | 6/162
Other Adverse Events (participants affected / at risk) | 0/170 | 0/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A TKA Without VERASENSE (N=170) | Group B TKA With VERASENSE (N=162)
Stiffness (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) — Stiffness causing in mobilization under anesthesia
Chest pain unspecific (General disorders) | 1 (1) | 0 (0)
Deep joint infection (Infections and infestations) | 0 (0) | 2 (2)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kidney injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The evaluation of tibiofemoral rotational alignment using intraoperative sensing which was highlighted in the study title, was identified off-label. Any data which should have been evaluated off-label are not included in the study results. Since the study has already ended at time point of data posting, the study title was not subsequently updated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT02286739/Prot_SAP_000.pdf